CLINICAL TRIAL: NCT03082469
Title: Pancreatitis CytoSorbents (CytoSorb®) Inflammatory Cytokine Removal: A Prospective Study.
Brief Title: Pancreatitis CytoSorbents (CytoSorb®) Inflammatory Cytokine Removal
Acronym: PACIFIC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: CytoSorbents Europe GmbH (Industry)
Responsible Party: Principal Investigator, Wolfgang Huber, Professor Dr. Wolfgang Huber, Technical University of Munich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACIFIC 10-2015
Record Dates: First submitted 2017-01-13; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Pancreatitis, Acute; SIRS
Keywords: Severe acute pancreatitis; Haemodynamic monitoring; Cytokine removal; Vasopressor dependency index
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: Inflammatory cytokine removal by Cyto Sorb treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CytoSorb (Active Comparator): CytoSorb therapy for 48h
  Interventions: Device: CytoSorb
- Matched controls (No Intervention): 60 matched controls with SAP and transpulmonary thermodilution monitoring

INTERVENTIONS:
Device: CytoSorb — Two consecutive 24h treatments with the CytoSorb-device
  Arms: CytoSorb

SUMMARY:
Severe acute pancreatitis (SAP) has a mortality of up to 42%. The outcome of SAP is related to the development of SIRS and consecutive organ failures. Due to the lack of a causative therapy except the removal of bile duct stones, therapy is predominantly symptomatic.

With regard to a marked inflammatory response ("cytokine storm") during the early phase of SAP extracorporeal cytokine removal is a promising therapeutic approach.

This prospective case control study investigates the impact of early extracorporeal cytokine adsorption with the CytoSorb®-device on haemodynamics (primary endpoint) and several secondary outcomes.

DETAILED DESCRIPTION:
Severe acute pancreatitis (SAP) has a mortality of up to 42%. The outcome of SAP is related to the development of SIRS and consecutive organ failures. Due to the lack of a causative therapy except the removal of bile duct stones, therapy is predominantly symptomatic.

Severity and mortality are associated to an early systemic inflammatory response syndrome (SIRS) and to septic complications at a later stage of disease.

With regard to a marked inflammatory response ("cytokine storm") during the early phase of SAP extracorporeal cytokine removal is a promising therapeutic approach.

This prospective case control study investigates the impact of early extracorporeal cytokine adsorption with the CytoSorb® device on haemodynamics (primary endpoint) and several secondary outcomes.

Patients with high probability of SAP (APACHE-II-score ≥10) are eligible for 7 days after the onset of pain.

The patients will be treated for 48h with two consecutive 24h sessions of cytokine absorption with the CytoSorb®-device.

All patients will be under haemodynamic Monitoring with transpulmonary thermodilution The primary endpoint is defined as an improvement of the vasopressor dependency index of ≥20% (if no vasoactive drugs are used at baseline, the cardiac power index cardiac power index (CPI) will be used as primary endpoint).

The outcome analysis will be based on comparison of the incidence of the primary endpoint in 30 Intervention patients compared to 60 matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Proven acute pancreatitis:

  * typical pain
  * at least 3-fold increase in serum lipase
  * onset of pain within 7 days before inclusion AND
* APACHE-II ≥10 AND
* ≥1 criterion of "severe sepsis" AND
* Haemodynamic monitoring with transpulmonary thermodilution AND
* ≥ 1 marker of poor prognosis of acute pancreatitis:

  * Haematocrit > 44% (men), >40% (women)
  * Blood glucose > 125 mg/dL
  * C-reactive protein (CRP) > 10mg/dL
  * Computed tomography score category C-E
  * Age >55 years
  * Leukocytes >16 G/L
  * Glutamate oxaloacetate transferase (GOT) >250 U/L
  * Lactate dehydrogenase (LDH) >350 U/L
  * Calcium <2,0mmol/L

Exclusion Criteria:

* pregnancy
* lack of informed consent of patient or representative
* pre-existing disease with life expectancy <3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-15 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Haemodynamics | Within 48h after the onset of CytoSorb treatment
  Improvement of the vasopressor dependency index >=20%. (Improvement of cardiac power index >=20% in case of no vasopressor use at baseline)

SECONDARY OUTCOMES:
Mortality-1 | 28 days from inclusion into the study
  28-days-mortality
Mortality-2 | From admission to the ICU until discharge or transfer from the ICU (up to one year)
  ICU-mortality
Mortality-3 | From admission to discharge from the hospital (up to one year)
  Hospital-mortality
Inflammation | Within 48h after the onset of CytoSorb treatment
  IL-6, CRP and PCT-values levels compared to before CytoSorb treatment
Respiratory outcome | Within 28 days after the onset of CytoSorb treatment
  Ventilator-free days
Renal function and its Change over time | Within 28 days after the onset of CytoSorb treatment
  Daily classification according to KDIGO; comparison vs. before Cyto Sorb treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Huber, Professor, Principal Investigator — II. Medizinische Klinik; Klinikum rechts der Isar; Technische Universität München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huber W, Algul H, Lahmer T, Mayr U, Lehmann M, Schmid RM, Faltlhauser A. Pancreatitis cytosorbents (CytoSorb) inflammatory cytokine removal: A Prospective Study (PACIFIC). Medicine (Baltimore). 2019 Jan;98(4):e13044. doi: 10.1097/MD.0000000000013044. PMID 30681551